CLINICAL TRIAL: NCT05053464
Title: Developing New Models of Care for People With Fibromyalgia: Designing a DCE to Understand Patients' Preferences for Alternative Models of Care
Brief Title: A DCE to Understand Patients' Preferences for Alternative Models of Care
Status: Completed | Type: Observational
Sponsor: University of Aberdeen (Other)
Responsible Party: Sponsor
Other Study IDs: 2-041-21
Record Dates: First submitted 2021-09-03; First posted 2021-09-22 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A pilot survey for a Discrete Choice Experience to understand the strength of patient's preferences for alternative models of care for fibromyalgia.

DETAILED DESCRIPTION:
We will use the Discrete Choice Experiment (DCE) method to elicit preferences for alternative models of care for people with fibromyalgia. The DCE is a choice-based survey that quantifies preferences for attributes (or features) of goods, services or policy interventions. It assumes that any good or service (in this case models of care for fibromyalgia) can be described by its attributes and the measure (or 'levels') of these attributes. Each respondent faces a series of hypothetical scenarios (choice sets) composed of two or more alternatives. In each choice set, respondents are asked to choose their preferred scenario. The principle underlying a DCE is choices are made based on the features (or attributes) of different actions. Therefore, a DCE enables researchers to gain insight into the relative importance of each attribute, and the trade-offs between attributes.

This study is a survey of participants identified from a previous study about chronic widespread pain ("MAintaining MusculOskeleTal Health" - MAmMOTH). As part of the MAmMOTH study, a randomly selected sample of adults aged 25 years and over registered with participating general practices in Scotland were mailed a screening questionnaire. All individuals who returned the completed screening questionnaire and who met some criteria for fibromyalgia and consented to be contacted for future health survey research were approached for a further survey, the DEHLTA study. The DEHLTA survey questionnaire asked participants if they had ever received a diagnosis of fibromyalgia. From respondents to the DEHLTA study, individuals who said they had a diagnosis of fibromyalgia and who consented to be contacted for future studies will be eligible to participate in the current pilot study. We estimate this will be approximately 80 individuals.

Inclusion criteria are:

* Reporting a diagnosis of fibromyalgia in the DEHLTA survey
* Consenting to be contacted for future health survey research in the DEHLTA survey

Exclusion criteria are:

* Not reporting a diagnosis of fibromyalgia in the DEHLTA survey
* Not consenting to be contacted for future health survey research in the DEHLTA survey

Eligible individuals will receive a one-off paper questionnaire (including an invitation letter, a patient information sheet, and a prepaid, preaddressed envelope) and be invited to participate in the current study. A reminder letter will be mailed two weeks later. Mailings will be carried out by study staff at the University of Aberdeen.

We will analyse the feasibility of the model of data collection and quality of the questionnaire responses by estimating response rate, questionnaire completion times, item response and qualitative feedback on question items. In addition, we will assess frequencies and associations in choice responses to examine the strength of preferences relating to service provision in terms of the specified attributes (time to diagnosis, diagnosis provider, treatment type, waiting time, and type of on-going help and support). The data analysis conducted will inform the design of a larger study involving participants from a national patient organisation.

ELIGIBILITY:
Inclusion Criteria:

* Reporting a diagnosis of fibromyalgia in the DEHLTA survey
* Consenting to be contacted for future health survey research in the DEHLTA survey

Exclusion Criteria:

* Not reporting a diagnosis of fibromyalgia in the DEHLTA survey
* Not consenting to be contacted for future health survey research in the DEHLTA survey

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Respondents to a previous survey questionnaire who had told us they had a diagnosis of fibromyalgia
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2021-08-25 (Actual); Primary Completion 2021-10-08 (Actual); Study Completion 2021-10-08 (Actual)

PRIMARY OUTCOMES:
Patient Preferences for treatment for fibromyalgia | The outcome will be measured at a single timepoint, i.e. the time of completion of the survey questionnaire. The survey will be carried out during August and September 2021.
  This will be derived from the participants' answers to discrete choice questions

CONTACTS AND LOCATIONS:
Locations (1):
- University of Aberdeen, Aberdeen, United Kingdom

IPD SHARING:
Plan to Share IPD: No